CLINICAL TRIAL: NCT00165217
Title: A Phase II Trial of Capecitabine and Thalidomide in Previously Treated Metastatic Colorectal Carcinoma
Brief Title: Capecitabine and Thalidomide in Previously Treated Metastatic Colorectal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-141
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Colorectal Adenocarcinoma
Keywords: capecitabine; thalidomide; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Thalidomide

INTERVENTIONS:
Drug: Capecitabine
Drug: Thalidomide

SUMMARY:
The purpose of this study is to collect information about the antitumor activity and the safety of capecitabine and thalidomide in patients with colorectal cancer.

DETAILED DESCRIPTION:
* Patients will take capecitabine orally twice a day for two weeks followed by a one week break period. These three week cycles will continue as long as the patient continues to benefit from the the therapy and does not experience intolerable side effects.
* Thalidomide will be taken orally once daily in the evening. Each week teh daily dose of the medication will be increased by 100mg as long as the patient is not experiencing any moderate to severe side effects. The dose will be increased in this manner until the daily dose is 600mg. If side effects do develop, the dose will either be held constant or decreased until the side effects resolve. If the side effects do not resolve, treatment will be stopped.
* Before starting treatment and periodically throughout the study, a physical exam, routine blood tests, scans and x-rays will be done to monitor the body's response to the treatment.
* For women patients, pregnancy tests will be performed every 3 weeks while on therapy.
* Scans and x-rays will be performed every 9 weeks (after every 3 cycles of treatment) to follow the effects of the study drugs on the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of colorectal adenocarcinoma with radiological or cytological evidence of stage IV (metastatic) disease
* Measurable tumor
* Serum creatinine < 1.5 mg/dl
* Total bilirubin < 2.0 mg/dl
* AST < 5 x ULN
* ANC > 1,500/mm3
* Platelets > 100,000/mm3
* Hemoglobin > 9.0 gm/dl
* Must have received at least one prior chemotherapy regimen for metastatic colorectal cancer. At least 3 weeks must have passed since the last chemotherapy treatment
* 18 years of age or older
* ECOG performance status of less than or equal to 2
* Life expectancy of greater than 12 weeks

Exclusion Criteria:

* Prior treatment with mitomycin C or nitrosourea compounds
* Prior treatment with capecitabine or thalidomide
* Clinically apparent central nervous system metastases or carcinomatous meningitis
* Peripheral neuropathy of grade 2 or greater severity
* Myocardial infarction in the past 6 months
* Major surgery in the past 2 weeks
* Uncontrolled serious medical or psychiatric illness
* Pregnant or lactating women
* Concurrent malignancy of any site, except limited basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Known allergy to 5-FU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37
Dates: Start 2001-11; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
To assess the anti-tumor activity of capecitabine and thalidomide when administered to patients with previously treated metastatic colorectal cancer.

SECONDARY OUTCOMES:
To evaluate the safety of capecitabine and thalidomide in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Fuchs, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts